CLINICAL TRIAL: NCT00716638
Title: Trauma-focused CBT vs. EMDR in the Treatment of Posttraumatic Stress Disorder
Brief Title: Trauma-focused CBT Versus EMDR in the Treatment of Posttraumatic Stress Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Paul M.G.Emmelkamp, Professor, VU University of Amsterdam
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2008-KP-343
Record Dates: First submitted 2008-07-14; First posted 2008-07-16 (Estimated); Last update posted 2018-09-13 (Actual); Status verified 2018-09

CONDITIONS: Stress Disorders, Post-Traumatic
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment group 1 (Experimental): Trauma-focused Cognitive Behavior Therapy (TF-CBT)
  Interventions: Behavioral: Trauma-focused Cognitive Behavior Therapy
- Treatment group 2 (Experimental): Eye Movement Desensitization and Reprocessing (EMDR)
  Interventions: Behavioral: Eye Movement Desensitization and Reprocessing (EMDR)

INTERVENTIONS:
Behavioral: Trauma-focused Cognitive Behavior Therapy — This intervention comprises 10 sessions of trauma-focused cognitive behavior therapy for PTSD with the components (a) prolonged imaginal exposure, (b) in vivo exposure, and (c) cognitive restructuring.
  Arms: Treatment group 1
Behavioral: Eye Movement Desensitization and Reprocessing (EMDR) — This intervention comprises 10 sessions of EMDR according to the standard protocol.
  Arms: Treatment group 2

SUMMARY:
This study will evaluate the effectiveness of trauma-focused cognitive behaviour therapy (TF-CBT) versus eye movement desensitization and reprocessing (EMDR) in the treatment of trauma survivors with post-traumatic stress disorder (PTSD). Patients will be randomly assigned to TF-CBT or EMDR. Follow-up assessments will be conducted at 3 and 12 months post-treatment. In addition to comparing the efficacy of the two protocols, an additional focus will lie on identifying predictors for treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* A full diagnosis of PTSD according to the DSM-IV or subthreshold PTSD (criteria for intrusive re-experiencing are fulfilled and either three avoidance/numbing symptoms or two hyperarousal symptoms are present)
* PTSD is related to one or more single-event traumas and participants have a clear memory of this event/these events (sufficient for constructing scenes to be used in exposure)
* Age between 18 and 70
* Sufficient fluency in Dutch to complete treatment and research protocol
* If participants are using anti-depressants, they need to be on a stable dose for at least 2 weeks before the beginning of treatment and remain on this dose throughout the treatment.

Exclusion Criteria:

* Dementia or other severe cognitive impairment
* Psychosis
* Depression with suicidal ideation
* Bipolar disorder
* Borderline Personality Disorder
* Anti-social personality disorder
* Substance dependence
* Current use of tranquilizers
* Exposure to prolonged and/or chronic trauma ("type-II-trauma")

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
PTSD symptom severity: (a) interviewer rating (PSS-I); (b) self-report (PDS) | Assessed at post-treatment, 3 months and 12 months follow-up

SECONDARY OUTCOMES:
Depressive symptom severity (Beck Depression Inventory, BDI) | assessed at post-treatment, 3 months and 12 months follow-up
Severity of anxiety symptoms (Beck Anxiety Inventory, BAI) | assessed at posttreatment, 3 months and 12 months follow-up
Trauma-related appraisal (Posttraumatic Cognitions Inventory, PTCI) | post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Paul MG Emmelkamp, Professor, Principal Investigator — University of Amsterdam; Thomas Ehring, PhD, Study Director — University of Amsterdam
Locations (1):
- PsyQ, Zaandam, Netherlands